CLINICAL TRIAL: NCT07195422
Title: Evaluation of the Japet.W+ Medical Device for Low Back Pain Management: Performance and Safety Analysis Across Two Patients' Groups
Brief Title: Evaluation of the Japet.W+ Medical Device for Low Back Pain Management
Acronym: EXODOMICILE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Japet Medical Devices (Industry)
Collaborators: University Hospital, Clermont-Ferrand (Other); Hôpital Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2024-A01665-42
Record Dates: First submitted 2025-01-03; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-01

CONDITIONS: Low Back Pain
Keywords: Low back pain; Active discopathy; Japet.W+; Medical device; Pain assessment; Quality of life
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Active Comparator): Period 1 (week 1-8): Current care / Washout period (week 9-10) / Period 2 (week 11-18): Current care + Japet.W+
  Interventions: Device: Japet.W+; Device: Control (Standard treatment)
- Group B (Active Comparator): Period 1 (week 1-8): Current care + Japet.W+ / Washout period (week 9-10) / Period 2 (week 11-18): Current care
  Interventions: Device: Japet.W+; Device: Control (Standard treatment)

INTERVENTIONS:
Device: Japet.W+ — Current care of low back pain and wearing the Japet.W+
  Other Names: Experimental
Device: Control (Standard treatment) — Current care of low back pain

SUMMARY:
The JAPET.W+ medical device is a new dynamic distraction support system. It could be considered as a new solution in the therapeutic arsenal for managing common low back pain. This study aims to assess the effectiveness of this device among the two targeted populations during daily use. Each patient will be asked to estimate the intensity of their low back pain several times during the clinical investigation. Our main hypothesis is a reduction in low back pain while wearing the device. The secondary hypothesis is a decrease in activity limitations, an increase in participation, an improvement in quality of life, and a reduction in healthcare product and medication consumption.

ELIGIBILITY:
Inclusion Criteria:

* Non-specific chronic low back pain with active discopathy OR Non-specific chronic low back pain without active discopathy,
* 18 years ≤ Age < 80 years,
* Average pain intensity (VAS) over the last week ≥ 40/100,
* Patient affiliated to the health social security system,
* Patient able to understand the information relating to the study and to sign the informed consent form.

Exclusion Criteria:

* Specific low back pain (infectious, inflammatory, tumorous, or traumatic in origin).
* Motor neurological deficits (peripheral or central).
* Extrapyramidal syndrome.
* Treatment with implanted neurostimulation.
* Severe heart or circulatory disease or respiratory problems.
* Arthrodesis or disc replacement.
* Surgery for herniated disc (<3 months).
* Spinal fracture or floating ribs (<3 months).
* Skin lesions on the trunk, history of contusions or skin lesions following traction of the trunk.
* Pregnancy.
* Patients who cannot tolerate the JAPET.W+ device during an initial trial.
* Patients under guardianship, curatorship, or legal protection.
* Participation in another clinical trial.
* Patients who have worn a device designed to reduce lower back pain regularly during the 2 weeks prior to inclusion (lumbar belt, corset, exoskeleton).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | Comparison of the difference Δ1=VASweek8 - VASweek1 and Δ2=VASweek18-VASweek11.
  Pain VAS is a unidimensional measure of pain intensity (from 0: no pain to 100: severe pain), used to record the progression of pain in patients or to compare the severity of pain between patients with similar conditions. The VAS has been widely used in various adult populations, for example people suffering from chronic low back pain.

SECONDARY OUTCOMES:
Adverse events | Week 4 day 7, Week 8 day 7, Week 14 day 7 and Week 18 day 7
Rate of device failure | Group B: Week 4 day 7, Week 8 day 7 / Group A: Week 14 day 7 and Week 18 day 7
Functional disability | Beginning and end of each period (Week 1 day 1, Week 8 day 7, Week 11 day 1, Week 18 day 7).
  Measurement of specific activity limitation using the Roland-Morris score
Quality of life | Beginning and end of each period (Week 1 day 1, Week 8 day 7, Week 11 day 1, Week 18 day 7).
  The SF-12 physical (PCS-12) and mental (MCS-12) component summary scales are scored using norm-based methods. Physical and mental regression weights and a constant for both measures come from the general U.S. population. Both the PCS-12 and MCS-12 scales are transformed to have a mean of 50 and a standard deviation of 10 in the general U.S. population.
  The minimum possible PCS score (standard version of the SF-12) is 9.9 points and the maximum is 76.0 points. For the MCS, the minimum is 3.2 and the maximum is 77.9. In both cases, the higher the score, the better the patient's health status.
Adherence to Japet.W+ | Recovery of Japet.W+ usage time after 28 days and 56 days of use. Group A (using the device during the second period): Week 14, day 7, and Week 18, day 7. Group B (using the device during the first period): Week 4, day 7, and Week 8, day 7.
  Recovery of Japet.W+ usage time.
Number of healthcare products consumed (drugs, medical appointments, physiotherapy sessions, etc.) | Information retrieved 3 times per period (D+7, D+28, D+56). Period 1: Week 1 day 7, Week 4 day 7, Week 8 day 7. Period 2: Week 11 day 7, Week 14 day 7, and Week 18 day 7.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital de Cochin, APHP, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided